CLINICAL TRIAL: NCT00671372
Title: A Phase Ib, Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of Multiple Doses of Dulanermin Administered Intravenously in Combination With Camptosar®/Erbitux® Chemotherapy or the Folfiri Regimen With or Without Bevacizumab in Subjects With Previously Treated Metastatic Colorectal Cancer
Brief Title: A Study of Dulanermin Administered in Combination With Camptosar®/Erbitux® Chemotherapy or FOLFIRI (With or Without Bevacizumab) in Subjects With Previously Treated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APO3583g; GO00933
Record Dates: First submitted 2008-04-18; First posted 2008-05-05 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
Keywords: CRC; Metastatic CRC; APO2L/TRAIL
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Cetuximab; TNFSF10 protein, human; Irinotecan

ARMS (2):
- Cohorts 1-5 (Experimental)
  Interventions: Drug: cetuximab; Drug: dulanermin; Drug: irinotecan
- Cohorts 6, 6A, 7, 7A (Experimental)
  Interventions: Drug: FOLFIRI regimen; Drug: bevacizumab; Drug: dulanermin

INTERVENTIONS:
Drug: FOLFIRI regimen — Intravenous repeating dose
  Arms: Cohorts 6, 6A, 7, 7A
Drug: bevacizumab — Intravenous repeating dose (for Cohort 6 subjects not previously treated with bevacizumab)
  Arms: Cohorts 6, 6A, 7, 7A
Drug: cetuximab — Intravenous repeating dose
  Arms: Cohorts 1-5
Drug: dulanermin — Intravenous repeating dose
Drug: irinotecan — Intravenous repeating dose
  Arms: Cohorts 1-5

SUMMARY:
This study will assess the safety and pharmacokinetics of adding dulanermin to Camptosar®/Erbitux® or the FOLFIRI regimen (Camptosar®, 5-FU, and leucovorin) plus bevacizumab (only for Cohort 6 subjects who have not received prior bevacizumab therapy).

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age >= 18 years
* Histologically confirmed CRC with evidence of metastases and measurable tumor lesion(s)
* Progression of disease following, or intolerance to, treatment with 5-fluorouracil-based therapy
* Progression of disease during or within =< 6 months following the last dose of a prior first-line treatment with a fluoropyrimidine and oxaliplatin-based chemotherapy plus bevacizumab for metastatic disease
* Use of an effective means of contraception for women of childbearing potential and men with partners of childbearing potential (use per institutional standard)
* Life expectancy of > 3 months
* Willingness and capability to be accessible for study follow-up

Exclusion Criteria:

* Prior radiotherapy to a measurable, metastatic lesion(s) to be used to measure response
* Radiation therapy to a peripheral lesion within 14 days prior to Day 1; Radiation therapy to a thoracic, abdominal or pelvic field within 28 days prior to Day 1
* Chemotherapy, hormonal therapy, or immunology within 4 weeks prior to Day 1
* Previous exposure to DR4-targeted therapy or DR5-targeted therapy
* Evidence of clinically detectable ascites on Day
* Other invasive malignancies within 5 years prior to Day 1 (other than basal cell carcinoma of the skin or in situ carcinoma of the cervix)
* History or evidence upon physical examination of CNS disease
* Active infection requiring parenteral antibiotics on Day 1
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study and fine needle aspirations within 7 days prior to Day 1
* Pregnancy or lactation
* Serious nonhealing wound, ulcer, or bone fracture
* Current or recent participation in another experimental drug study
* Clinically significant cardiovascular disease
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk from treatment complications
* Cohort 5 only: Subjects who have a Kras mutation will be excluded from enrollment
* The following exclusion criteria apply only to subjects who have received prior bevacizumab and are enrolled in Cohort 6: four or more prior doses of bevacizumab therapy, inadequately controlled hypertension, history of hypertensive crisis or hypertensive encephalopathy, history of arterial thromboembolic event 6 months prior to Day 1, proteinuria, history of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of dulanermin administered in combination with Camptosar and Erbitux | Length of study
The safety and tolerability of dulanermin administered in combination with FOLFIRI (with or without Bevacizumab) | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Chia Portera, M.D., Study Director — Genentech, Inc.
Locations (10):
- United States (10):
  - Los Angeles, California
  - Redlands, California
  - San Francisco, California
  - Fort Myers, Florida
  - Harvey, Illinois
  - Buffalo, New York
  - Durham, North Carolina
  - Hershey, Pennsylvania
  - Nashville, Tennessee
  - Tacoma, Washington